CLINICAL TRIAL: NCT04324827
Title: Investigation of the Acute Effect of Myofascial Release Techniques and Dynamic Stretch on Vertical Jump Performance in Recreationally Active Individuals
Brief Title: Investigation of the Acute Effect of Myofascial Release Techniques and Dynamic Stretch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Principal Investigator, Bahçeşehir University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Jump.2019-07.19
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Graston Technique®, Dynamic Stretching, Foam Roller, Jumping Performance, Soft Tissue Mobilization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: There was a blind assessor (Physical Therapist) and completed the Optojump testing. Participants are also blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Graston Technique® Group (Experimental): The application was applied by a GT® certified therapist with 12 years of experience in orthopedic rehabilitation and soft tissue treatments. Hamstring, gastrosoleus and plantar fascia were scanned with GT® instruments and the treated soft tissue was treated. The instruments used differ according to the application protocol and regions are determined with reference to the GT® manual. The treatment lasted 8 minutes for each leg and was applied to both legs equally and by the same person for a total of 16 minutes.
  Interventions: Device: Graston Technique
- Foam Roller Group (Experimental): FR was applied to gastrosoleus and hamstring muscle groups and plantar fascia. TriggerPoint Grid X Foam Roller and Nano Foot X Roller were used in the application. Hamstring, gastrosoleus and plantar fascia for 3 minutes were performed for a single leg. The treatment lasted 8 minutes on one leg and was applied equally to both legs for a total of 16 minutes. Before the application, the participants were informed with verbal and visual warnings about how to do the applications. During the application, the participant was instructed about the time with a stopwatch. The patient himself regulated the pressure applied to the FR; however, the participant was instructed to apply FR as much body weight as possible. The frequency of application was about 0.5 Hz (ie, each rolling cycle lasted for about 2 seconds).
  Interventions: Device: Graston Technique
- Dynamic Stretch (Experimental): DS protocol was prepared with reference to the work of Faigenbaum et al 2005. The protocol consists of 10 dynamic exercises of 10 minutes of medium and high intensity. Each dynamic stretching exercise was performed at a distance of 13 meters. The participants were given a 10-second rest period between each exercise. The participants were given verbal feedback about their postures during the exercises and the video of the exercises was shown to the participant.
  Interventions: Other: Dynamic stretch exercise

INTERVENTIONS:
Device: Graston Technique — FR is a dense foam cylinder that the person rolls before using the body weight to warm up and increase their ROM. There are different types that vary in size, shape and density.
  Other Names: Foam Roller
  Arms: Foam Roller Group; Graston Technique® Group
Other: Dynamic stretch exercise — Dynamic stretch includes controlled movements in the active ROM for a joint. This type of exercise is actually the basis of sports movements used in training or competition.
  Arms: Dynamic Stretch

SUMMARY:
Fascia is a connective tissue that contains a large amount of water and contains blood vessels, nerves that surround the muscles and connect the various structures of the body. In the event of an injury, the fascia has to cause some limitations to reduce muscle spasms, neuromuscular changes and pain. In order to achieve this, it can adhere to muscles and other body structures. In the physically active population, these facial adhesions may cause a decrease in performance over time, while the body heals itself after mechanical stresses and injuries. It is remarkable that various facial techniques are tried and compared with each other in order to increase performance. The most noteworthy of these techniques is foam roller (FR) and instrument-assisted soft tissue mobilization (IASTM). As well as myofascial techniques, a preferred and highly studied method for performance improvement, especially before competitions, is dynamic stretching. The aim of this study is to compare the effects of these three techniques on vertical jump performance and their advantages over each other.

DETAILED DESCRIPTION:
Fascia is a connective tissue that contains a large amount of water and contains blood vessels, nerves that surround the muscles and connect the various structures of the body. In the event of an injury, the fascia has to cause some limitations to reduce muscle spasms, neuromuscular changes and pain. In order to achieve this, it can adhere to muscles and other body structures. In the physically active population, these facial adhesions may cause a decrease in performance over time, while the body heals itself after mechanical stresses and injuries. It is remarkable that various facial techniques are tried and compared with each other in order to increase performance. The most noteworthy of these techniques is foam roller (FR) and instrument-assisted soft tissue mobilization (IASTM).

The IASTM technique is a therapeutic approach developed by James Cyriax. There are many different instruments used for myofascial release. The most popular one is Graston Technique® (GT® ). With specially designed instruments, longitudinal pressure is applied along the fibers of the respective muscles. Damaged tissues are detected by varying tissue vibration under the instrument. The therapeutic efficacy of the instruments, in particular by microtrauma created in the damaged areas, induces local inflammation response, enhances scar tissue destruction, enhances adhesion relaxation, enhances collagen synthesis and stimulates connective tissue remodeling. In addition to its rehabilitative use, IASTM has been found to be effective as a method that stimulates the nerves in muscles and increases muscle strength, performance and endurance. In addition, as tissue mobility and range of motion increase, performance increases and shortening of the recovery period after physical activity occurs.

In addition to manual therapy methods for myofascial release techniques, there are also applications that patients can perform on their own. FR and Stick Roller are examples. The use of pre-competition FR increases joint range of motion, reduces pain and tension, increases blood flow and joint flexibility, and reduces injury rate when exercising. It also relaxes scar tissue and facial adhesions, regulates muscle tone, provides relaxation in excessively active muscles and improves movement quality.

FR application is carried out with a foam roller which can vary in size, shape and density. It has become popular in clinics and athletic training halls because of their ease of use and versatility. They are available in different lengths, making them easier to move and easier to maneuver in different parts of the body. Best used in the treatment of large muscle groups. Each muscle group has a defined position and protocol with different starting and ending points. Individuals with poor collagen load ability and individuals new to FR studies often have to spend more time on the cylinder to achieve the best results. Foam roller sessions can be held once or twice a day and can be used as a warm-up tool before a training session or as a regeneration option after training. It increases tissue extensibility by opening both IASTM and FR adhesions.

A preferred and highly studied method for performance improvement, especially before competitions, is dynamic stretching. Dynamic stretching (DS) exercises are used for warm-up and relaxation before and after sports exercises. It is one of the common applications used for preparation before physical exercise. Dynamic stretching exercises are a series of exercises to prepare the muscles and joints in the body for the activity to be done, to reduce the incidence of possible injuries and to accelerate the regeneration process after sports. In addition, there are studies showing that dynamic stretching exercises affect performance positively and it has been found to give better results in areas such as jump and sprint compared to static stretching exercises.

The aim of this study is to compare the effects of these three techniques on vertical jump performance and their advantages over each other.

ELIGIBILITY:
Inclusion Criteria:

* being between18-35 years old,
* being recreationally active,
* volunteering to participate in the study
* no pain complaints.

Exclusion Criteria:

* body mass index of 30 kg / m² or more,
* previous lower extremity surgery and joint,
* meniscus or ligament injury,
* chronic knee instability,
* cardiac, musculoskeletal, vestibular and neurological problems,
* long-term use of corticosteroids
* pregnancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-11-24 (Actual)

PRIMARY OUTCOMES:
The Optojump system (Microgate, Bolzano, Italy) | Pre evaluation before the intervention
  Vertical Jump Performance evaluation with The countermovement jump without armswing test
The Optojump system (Microgate, Bolzano, Italy) | post evaluation right after the intervention.
  Vertical Jump Performance evaluation with The countermovement jump without armswing test

CONTACTS AND LOCATIONS:
Overall Officials: Mert Batuhan Ekiz, PT, Study Chair — Bahçeşehir University Health Sciences Faculty; İlhan Can Kulak, PT, Study Chair — Bahçeşehir University Health Sciences Faculty
Locations (1):
- Pelin Pişirici, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided